CLINICAL TRIAL: NCT01522183
Title: An Observational, Non-Interventional, Multi-Center, Multi-National Study of Patients With Atypical Hemolytic-Uremic Syndrome (aHUS Registry)
Brief Title: Atypical Hemolytic-Uremic Syndrome (aHUS) Registry
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Other Study IDs: M11-001
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Atypical Hemolytic-Uremic Syndrome
Keywords: Atypical Hemolytic-Uremic Syndrome; aHUS; Thrombotic Microangiopathy; TMA
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-marketing safety data on patients treated and untreated with eculizumab or ravulizumab.

DETAILED DESCRIPTION:
The study will capture post-marketing safety data on patients treated with eculizumab or ravulizumab. Additionally, the study will collect information on the progression of disease in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any age, including minors, who have been diagnosed with aHUS
* Patients with or without an identified complement pathogenic variant or anti-complement factor antibody
* Able to give written informed consent. Patient or patient's parent/legal guardian must be willing and able to given written informed consent and the patient (if minor) must be willing to give written informed assent [if applicable as determined by the central Institutional Review Boards/Independent Ethics Committees (IRB/IEC)].
* ADAMTS13 > 5%, if performed.

Exclusion Criteria:

* Hemolytic Uremic Syndrome (HUS) only due to Shiga Toxin producing Escherichia coli (STEC).
* Unable to give written informed consent. Patient or patient's parent/legal guardian unable to give written informed consent. Patient (if minor) unable to give written informed assent (if applicable as determined by the central Institutional Review Boards/Independent Ethics Committees [IRB/IEC]).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients of any age, including minors, who have been diagnosed with aHUS; clinical diagnosis of aHUS, patients with or without an identified complement regulatory factor genetic abnormality or anti-complement factor antibody, ADAMTS13 > 5% (if performed)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-03-18 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who experience specified events | 10 years
  To collect and evaluate safety and effectiveness data specific to the use of eculizumab or ravulizumab in aHUS patients.
Time to first and subsequent occurrence of specified events. | 5 years
  To assess the long term manifestations of thrombotic microangiopathy (TMA) complications of aHUS as well as other clinical outcomes, including morbidity and mortality in aHUS patients, receiving eculizumab or ravulizumab treatment or other disease management approaches

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Saval, Study Director — Alexion Pharmaceuticals, Inc.
Locations (132):
- United States (9):
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Gainesville, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Columbus, Ohio
- Australia (10):
  - Clinical Trial Site 1, Westmead, New South Wales
  - Clinical Trial Site 2, Westmead, New South Wales
  - Clinical Trial Site, Cairns, Queensland
  - Clinical Trial Site, Herston, Queensland
  - Clinical Trial Site, Woolloongabba, Queensland
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Heidelberg, Victoria
  - Clinical Trial Site, Parkville, Victoria
  - Clinical Trial Site, Murdoch, Western Australia
  - Clinical Trial Site, Nedlands, Western Australia
- Belgium (10):
  - Clinical Trial Site, Brussels
  - Clinical Trial Site (Adult), Edegem
  - Clinical Trial Site (Pediatric), Edegem
  - Clinical Trial Site (pediatric), Ghent
  - Clinical Trial Site (Adult), Leuven
  - Clinical Trial Site (pediatric), Leuven
  - Clinical Trial Site (Adult), Liège
  - Clinical Trial Site (pediatric), Liège
  - Clinical Trial Site (adult), Woluwe-Saint-Lambert
  - Clinical Trial Site (Pediatric), Woluwe-Saint-Lambert
- Canada (4):
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
  - Clinical Trial Site, Québec, Quebec
- Clinical Trial Site, Odense, Denmark
- France (38):
  - Clinical Trial Site 1, Amiens
  - Clinical Trial Site 2, Amiens
  - Clinical Trial Site, Angers
  - Clinical Trial Site, Bayonne
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Brest
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Caen
  - Clinical Trial Site, Chambéry
  - Clinical Trial Site, Clermont-Ferrand
  - Clinical Trial Site, Dijon
  - Clinical Trial Site, Grenoble
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Montpellier
  - Clinical Trial Site 1, Nancy
  - Clinical Trial Site, Nancy
  - Clinical Trial Site, Nantes
  - Clinical Trial Site 1, Nantes
  - Clinical Trial Site, Nice
  - Clinical Trial Site 2, Paris
  - Clinical Trial Site 4, Paris
  - Clinical Trial Site 1, Paris
  - Clinical Trial Site 5, Paris
  - Clinical Trial Site 3, Paris
  - Clinical Trial Site, Perpignan
  - Clinical Trial Site, Poitiers
  - Clinical Trial Site, Pontoise
  - Clinical Trial Site, Rennes
  - Clinical Trial Site 1, Rouen
  - Clinical Trial Site 2, Rouen
  - Clinical Trial Site 1, Strasbourg
  - Clinical Trial Site 2, Strasbourg
  - Clinical Trial Site, Toulouse
  - Clinical Trial Site, Tours
  - Clinical Trial Site, Valenciennes
- Germany (7):
  - Clinical Trial Site, Essen
  - Clinical Trial Site 1, Hanover
  - Clinical Trial Site 2, Hanover
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Lübeck
  - Clinical Trial Site, Münster
  - Clinical Trial Site, Tübingen
- Clinical Trial Site, Beersheba, Israel
- Italy (9):
  - Clinical Trial Site 1, Bari
  - Clinical Trial Site 2, Bari
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Genova
  - Clinical Trial Site 1, Milan
  - Clinical Trial Site 2, Milan
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Roma
  - Clinical Trial Site, Torino
- Clinical Trial Site, Lodz, Poland
- Russia (3):
  - Clinical Trial Site 1, Moscow
  - Clinical Trial Site 2, Moscow
  - Clinical Trial Site, Saint Petersburg
- South Korea (18):
  - Clinical Trial Site, Dongan, Chungcheongnam-do
  - Clinical Trial Site, Seoul, Dongnam-ro
  - Clinical Trial Site, Anyang-si, Gyeonggi-do
  - Clinical Trial Site, Goyang-si, Gyeonggi-do
  - Clinical Trial Site, Daegu, Hyeonchung-ro
  - Clinical Trial Site, Gwangju, Jebong Ro
  - Clinical Trial Site, Daegu
  - Clinical Trial Site 1, Gyeonggi-do
  - Clinical Trial Site 2, Gyeonggi-do
  - Clinical Trial Site, Jeju-do
  - Clinical Trial Site, Jeollabuk-do
  - Clinical Trial Site 2, Seoul
  - Clinical Trial Site 3, Seoul
  - Clinical Trial Site 5, Seoul
  - Clinical Trial Site 6, Seoul
  - Clinical Trial Site 7, Seoul
  - Clinical Trial Site 4, Seoul
  - Clinical Trial Site 1, Seoul
- Spain (4):
  - Clinical Trial Site 1, Barcelona
  - Clinical Trial Site 2, Barcelona
  - Clinical Trial Site, Pamplona
  - Clinical Trial Site, Seville
- Switzerland (3):
  - Clinical Trial Site, Basel
  - Clinical Trial Site, Bern
  - Clinical Trial Site, Surich
- Taiwan (4):
  - Clinical Trial Site, Kaohsiung City
  - Clinical Trial Site, New Taipei City
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Taoyuan District
- Turkey (Türkiye) (3):
  - Clinical Trial Site, Ankara
  - Clinical Trial Site, Istanbul
  - Clinical Trial Site, Kayseri
- United Kingdom (7):
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, Exeter
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Newcastle
  - Clinical Trial Site, Southampton
  - Clinical Trial Site, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaeckler A, Al-Dakkak I, Saval N, Dieperink HH, Eygenraam M, Greenbaum LA, Isbel N, Walle JV. Effectiveness and Safety of Switching to Ravulizumab From Eculizumab in Kidney Transplant Recipients With Atypical Hemolytic Uremic Syndrome: A Global aHUS Registry Analysis. Clin Transplant. 2025 Sep;39(9):e70278. doi: 10.1111/ctr.70278. PMID 40875209
- [Derived] Halimi JM, Al-Dakkak I, Anokhina K, Ardissino G, Licht C, Lim WH, Massart A, Schaefer F, Walle JV, Rondeau E. Clinical characteristics and outcomes of a patient population with atypical hemolytic uremic syndrome and malignant hypertension: analysis from the Global aHUS registry. J Nephrol. 2023 Apr;36(3):817-828. doi: 10.1007/s40620-022-01465-z. Epub 2022 Sep 24. PMID 36152218
- [Derived] Woodward L, Johnson S, Walle JV, Beck J, Gasteyger C, Licht C, Ariceta G; aHUS Registry SAB. An innovative and collaborative partnership between patients with rare disease and industry-supported registries: the Global aHUS Registry. Orphanet J Rare Dis. 2016 Nov 21;11(1):154. doi: 10.1186/s13023-016-0537-5. PMID 27871301
- [Derived] Licht C, Ardissino G, Ariceta G, Cohen D, Cole JA, Gasteyger C, Greenbaum LA, Johnson S, Ogawa M, Schaefer F, Vande Walle J, Fremeaux-Bacchi V. The global aHUS registry: methodology and initial patient characteristics. BMC Nephrol. 2015 Dec 10;16:207. doi: 10.1186/s12882-015-0195-1. PMID 26654630
- [Derived] Belingheri M, Possenti I, Tel F, Paglialonga F, Testa S, Salardi S, Ardissino G. Cryptic activity of atypical hemolytic uremic syndrome and eculizumab treatment. Pediatrics. 2014 Jun;133(6):e1769-71. doi: 10.1542/peds.2013-2921. Epub 2014 May 19. PMID 24843058
- [Derived] Ardissino G, Possenti I, Tel F, Testa S, Paglialonga F. Time to change the definition of hemolytic uremic syndrome. Eur J Intern Med. 2014 Feb;25(2):e29. doi: 10.1016/j.ejim.2013.12.002. Epub 2013 Dec 21. No abstract available. PMID 24360866